CLINICAL TRIAL: NCT01317849
Title: Folic Acid and B Vitamins for Secondary Prevention of Stroke : A Double-blinded Randomized Controlled Trial
Brief Title: China Stroke Secondary Prevention Trial
Acronym: CSSPT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: financial assistance financial assistance financial assistance financial assistance financial assistance without financial assistance
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: xijing-003
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: folic acid; B vitamins; secondary prevention; stroke; randomized controlled trial; homocysteine
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Folic Acid; Vitamin B 6; Pyridoxine; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin supplements (Experimental)
  Interventions: Drug: Folic Acid; Drug: Vitamin B6; Drug: Vitamin B12
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Folic Acid — 0.8mg
  Other Names: folate
  Arms: vitamin supplements
Drug: Vitamin B6 — 10mg
  Other Names: Pyridoxine
  Arms: vitamin supplements
Drug: Vitamin B12 — 500ug
  Other Names: Cyanocobalamin
  Arms: vitamin supplements
Drug: placebo — 0.8 mg
  Arms: Placebo
Drug: placebo — 10mg
  Arms: Placebo
Drug: placebo — 500ug
  Arms: Placebo

SUMMARY:
The CSSPT study is a multi-center, randomized, double blinded, placebo-controlled secondary stroke prevention trial in China to determine whether the addition of folic acid and vitamin supplements will reduce recurrent stroke events and other combined incidence of recurrent vascular events and vascular death.

DETAILED DESCRIPTION:
The CSSPT study is a multi-center, randomized, double blinded, placebo-controlled secondary stroke prevention trial in China to determine whether the addition of folic acid and vitamin supplements will reduce recurrent stroke events and other combined incidence of recurrent vascular events and vascular death in patients with recent stroke or transient ischemic attack (TIA). All patients presenting to one of the participating neurologists or general physicians within one months of stroke (ischemic or hemorrhagic) or TIA (eye or brain) are eligible for this trial. Eligible patients will be randomized in a double-blinded fashion to receive multi-vitamins or placebo. The primary outcome event is the composite event "stroke, myocardial infarction, or death from any vascular cause", whichever occurs first. Our target is to recruit a total of 8,000 patients over the two years with a median follow-up of 3 years. Recruitment to the trial began in July 2011 and is planned to continue until December 2013. The investigators aim to complete final follow-up by the end of 2016.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting within one months of ischemic stroke (ischemic or hemorrhagic) or TIA
* Homocysteine level ≥ 15μmol／L
* Agree to take study medication;Be geographically accessible for follow-up
* Provide written informed consent

Exclusion Criteria:

* Other cause of ischemic stroke (cardioembolism; stroke of other determined etiology, and stroke of undetermined etiology according to TOAST subtypes) or hemorrhagic stroke (intracranial vascular malformations; cerebral amyloid angiopathy; trauma and bleeding disorders etc)
* Use of vitamin supplements containing folate, B6 or B12
* Pregnancy or women of child-bearing potential who are at risk of pregnancy
* Limited life expectancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Recurrent stroke | 3 years
Myocardial infarction | 3 years
Death due to other vascular causes | 3 years

SECONDARY OUTCOMES:
TIA | 3 years
Revascularization procedures | 3 years
Dementia | 3 years
Depression | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, MD, Study Director — the Department of Neurology , Xijing Hospital
Locations (1):
- Xijing Hosptial, Xi’an, Shanxi, China

REFERENCES:
- [Background] Liu X, Shi M, Xia F, Han J, Liu Z, Wang B, Yang F, Li L, Wu S, Wang L, Liu N, Lv Y, Zhao G. The China Stroke Secondary Prevention Trial (CSSPT) protocol: a double-blinded, randomized, controlled trial of combined folic acid and B vitamins for secondary prevention of stroke. Int J Stroke. 2015 Feb;10(2):264-8. doi: 10.1111/ijs.12017. Epub 2013 Mar 12. PMID 23490255